CLINICAL TRIAL: NCT06077773
Title: Phase 2, Multicenter, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Effects of EP262 in Subjects With Chronic Spontaneous Urticaria (CALM-CSU)
Brief Title: Phase 2, Multicenter, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Effects of EP262 in Subjects With Chronic Spontaneous Urticaria
Acronym: CALM-CSU
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Strategic Business Decision
Sponsor: Escient Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EP-262-201
Record Dates: First submitted 2023-10-05; First posted 2023-10-11 (Actual); Results first posted 2025-12-05 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-11

CONDITIONS: Chronic Spontaneous Urticaria
Keywords: Chronic Spontaneous Urticaria; Chronic Urticaria; Urticaria; EP262; CALM-CSU; CALM
MeSH Terms: conditions — Chronic Urticaria; Urticaria

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- EP262 50 mg (Experimental)
  Interventions: Drug: Oral EP262
- EP262 150 mg (Experimental)
  Interventions: Drug: Oral EP262
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- EP262 25 mg (Experimental)
  Interventions: Drug: Oral EP262

INTERVENTIONS:
Drug: Oral EP262 — Once daily
  Arms: EP262 150 mg; EP262 25 mg; EP262 50 mg
Drug: Placebo — Once daily
  Arms: Placebo

SUMMARY:
Phase 2, Multicenter, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Effects of EP262 in Subjects with Chronic Spontaneous Urticaria

ELIGIBILITY:
Inclusion Criteria:

* Documented history of chronic spontaneous urticaria (CSU) with a UAS7 greater than or equal to 16 despite stable treatment with H1 antihistamine consistent with standard of care
* Must be on a stable dose of H1 antihistamine up to 4 times the approved dose per local treatment guidelines

Exclusion Criteria:

* Urticaria with a clear underlying etiology other than CSU
* Urticaria with a clearly defined or sole trigger (chronic inducible urticaria)
* Other active skin diseases associated with chronic pruritus (eg, atopic dermatitis, bullous pemphigoid, prurigo nodularis, dermatitis herpetiformis)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2023-09-25 (Actual); Primary Completion 2024-12-18 (Actual); Study Completion 2025-01-16 (Actual)

CONTACTS AND LOCATIONS:
Locations (48):
- United States (34):
  - AllerVie Clinical Research, Birmingham, Alabama
  - Scottsdale Clinical Trials, Scottsdale, Arizona
  - Little Rock Allergy & Asthma Clinical Research Center, Little Rock, Arkansas
  - First OC Dermatology Research, Inc., Fountain Valley, California
  - Allergy and Asthma Specialists Medical Group, Huntington Beach, California
  - Antelope Valley Clinical Trials, Los Angeles, California
  - Allervie Clinical Research, Destin, Florida
  - University of Miami Itch Center, Miami, Florida
  - Florida Center for Allergy and Asthma Research, Miami, Florida
  - NuLine Clinical Trial Center, Pompano Beach, Florida
  - Advanced Clinical Research Institute, Tampa, Florida
  - University of South Florida, Tampa, Florida
  - Treasure Valley Medical Research, Boise, Idaho
  - Dawes Fretzin Clinical Research Group, LLC, Indianapolis, Indiana
  - Southern Indiana Clinical Trials, New Albany, Indiana
  - The Indiana Clinical Trials Center, Plainfield, Indiana
  - Velocity Clinical Research, Overland Park, KC Asthma & Allergy, Overland Park, Kansas
  - Allergy & Asthma Specialists, P.S.C., Owensboro, Kentucky
  - Johns Hopkins University, Baltimore, Maryland
  - Chesapeake Clinical Research, Inc., White Marsh, Maryland
  - The Clinical Research Center LLC, St Louis, Missouri
  - Montana Medical Research, Inc., Missoula, Montana
  - Las Vegas Clinical Trials, North Las Vegas, Nevada
  - Corning Center for Clinical Research, Horseheads, New York
  - Bobby Buka MD, PC, New York, New York
  - Allergy Partners Clinical Research, Asheville, North Carolina
  - Bernstein Clinical Research Center, LLC, Cincinnati, Ohio
  - Toledo Institute of Clinical Research Inc., Toledo, Ohio
  - Vital Prospects Clinical Research Institute, PC, Tulsa, Oklahoma
  - Allergy and Clinical Immunology Associates, Pittsburgh, Pennsylvania
  - Clinical Partners, LLC, Johnston, Rhode Island
  - National Allergy and Asthma Research, LLC., North Charleston, South Carolina
  - Progressive Clinical Research, PA, San Antonio, Texas
  - Allergy Associates of Utah, Murray, Utah
- Canada (3):
  - Red Maple Trials Inc., Ottawa, Ontario
  - Evidence Based Medical Educator Inc, Toronto, Ontario
  - Centre de Recherche Saint-Louis, Québec, Quebec
- Germany (4):
  - Medizinische Hochschule Hannover, Hanover, Lower Saxony
  - Universitatsmedizin Mainz der Johannes Gutenberg-Universitat, Mainz, Rhineland-Palatinate
  - Universitätsklinikum Carl Gustav Carus an der Technischen Universität Dresden, Dresden, Saxony
  - Institut fur Allergieforschung Charite - Universitatsmedizin Berlin, Berlin
- Centre for Human Drug Research, Leiden, South Holland, Netherlands
- Poland (3):
  - Prywatna Praktyka Lekarska Ewa Ring, Warsaw, Masovian Voivodeship
  - Pim Mswia, Warsaw, Masovian Voivodeship
  - Centrum Badan Klinicznych PI-House Sp. z o.o., Gdansk, Pomeranian Voivodeship
- Spain (3):
  - Hospital del Mar, Barcelona
  - Hospital Clinico San Carlos, Madrid
  - Hospital Arnau de Vilanova, Valencia

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study was conducted at 33 study sites in the United States, Germany, Canada, Poland, Spain, and the Netherlands. The study was terminated following the completion of Part 1 due to business reasons; Part 2 was not enrolled.
Groups:
- Placebo: Participants received matching placebo once daily for 6 weeks.
- EP262 50 mg: Participants received oral EP262 50 milligrams (mg) once daily for 6 weeks.
- EP262 150 mg: Participants received oral EP262 150 mg once daily for 6 weeks.
Period: Overall Study
Arm/Group | Placebo | EP262 50 mg | EP262 150 mg
Started | 38 | 37 | 38
Completed | 37 | 36 | 35
Not Completed | 1 | 1 | 3
Not completed — Withdrawal by Subject | 1 | 0 | 1
Not completed — Lost to Follow-up | 0 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | EP262 50 mg | EP262 150 mg | Total
Number analyzed (Participants) | 38 | 37 | 38 | 113
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.8 (16.1) | 43.6 (14.2) | 45.4 (14.6) | 44.6 (14.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 31 | 34 | 98
  Male | 5 | 6 | 4 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 6 | 5 | 16
  Not Hispanic or Latino | 33 | 31 | 33 | 97
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 32 | 25 | 25 | 82
  Black or African American | 4 | 9 | 8 | 21
  Asian | 0 | 1 | 4 | 5
  Brazilian | 0 | 0 | 1 | 1
  Not Reported | 0 | 1 | 0 | 1
  American Indian or Alaska Native/Black or African American/White | 1 | 0 | 0 | 1
  American Indian or Alaska Native/White | 1 | 0 | 0 | 1
  Middle Eastern | 0 | 1 | 0 | 1
Urticaria Activity Score over a 7-day period [Mean (Standard Deviation); unit: scores on a scale] — The UAS is a 24-hour self-evaluation based on the assessment of itch intensity and number of wheals. The UAS scales for itch (Itch Severity Score [ISS]) and wheal assessment (Hive Intensity Score [HSS]) are recorded as a score from 0 (no itch/hives) to 3 (intense itch/hives). ISS and HSS scores are summed over 7 consecutive days to create the ISS7 and HSS7 scores, which range from 0 to 21. The UAS score is the sum of the ISS and HSS scores. Daily UAS scores are summed over 7 consecutive days to create the UAS7 score, which ranges from 0 to 42. Higher scores indicate greater disease severity.
  scores on a scale | 29.52 (8.081) | 25.88 (7.129) | 25.95 (8.399) | 27.13 (8.009)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Visit 4 (Week 6) in the Urticaria Activity Score Over a 7-day Period (UAS7)
Description: The UAS is a chronic spontaneous urticaria (CSU)-specific, 24-hour self-evaluation, patient-reported outcome measure based on the assessment of key CSU symptoms: intensity of itch (assessed as the Itch Severity Score [ISS]) and number of wheals (assessed as the Hive Severity Score [HSS]). The UAS scales for both itch and wheal assessment are recorded as a score from 0 to 3, with 0 representing no itch/hives to 3 representing intense itch/hives. ISS and HSS scores are summed over 7 consecutive days to create the ISS7 and HSS7 scores, which range from 0 to 21. Higher scores indicate greater disease severity. The UAS score is the sum of the ISS and HSS scores. Daily UAS scores are summed over 7 consecutive days to create the UAS7 score, which ranges from 0 to 42. Higher scores indicate greater disease severity. The 7 daily UAS/ISS/HSS scores prior to or on the nominal Visit 4 (Week 6) date (including the nominal Week 6 visit date UAS/ISS/HSS score) were summed.
Time Frame: Baseline; Week 6
Population: Full Analysis Set: all randomized participants who took ≥1 dose of randomized study drug. Participants were analyzed according to randomized treatment assignment. Only participants with available data were analyzed. Mixed model for repeated measures (MMRM) included fixed effects for treatment group, week, treatment group by week interaction, prior omalizumab use, and the Baseline score as a covariate. Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | EP262 50 mg | EP262 150 mg
Number analyzed (Participants) | 35 | 36 | 34
scores on a scale | -10.41 (1.863) | -8.43 (1.844) | -11.95 (1.827)
Statistical Analysis 1: Comparison: Placebo vs EP262 50 mg; Test type: Superiority; p = 0.4059, MMRM — MMRM=mixed effects model for repeated measures; The p-value was based on the treatment group by week interaction term for the visit of interest; Least Square Mean Difference (LSMD) = 1.99, 90% CI 2-sided [-1.96 to 5.94], Standard Error of Mean 2.380 — LSMD = EP262 minus placebo
Statistical Analysis 2: Comparison: Placebo vs EP262 150 mg; Test type: Superiority; p = 0.5213, MMRM — The p-value was based on the treatment group by week interaction term for the visit of interest; LSMD = -1.53, 90% CI 2-sided [-5.49 to 2.42], Standard Error of Mean 2.385 — LSMD = EP262 minus placebo

2. Secondary Outcome: Number of Participants With Any Treatment-emergent Adverse Event (TEAE)
Description: An adverse event (AE) was defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. An AE could therefore have been any unfavorable or unintended sign (including a clinically significant abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product. Medical conditions present at baseline that worsened in severity or frequency after exposure to study drug were considered TEAEs. A TEAE was any condition that was not present prior to treatment with the study drug but appeared following treatment, was present at treatment initiation but worsened during treatment, or was present at treatment initiation but resolved and then reappeared while the individual was on treatment (regardless of the intensity of the AE when the treatment was initiated).
Time Frame: up to 81 days
Population: Safety Analysis Set: all participants who were randomized and took at least 1 dose of randomized study drug. Safety analyses were based upon treatment actually received.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | EP262 50 mg | EP262 150 mg
Number analyzed (Participants) | 38 | 37 | 38
Participants | 12 | 15 | 19

3. Secondary Outcome: Number of Participants With Any ≥Grade 3 TEAE
Description: An AE was any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. An AE could therefore have been any unfavorable or unintended sign (including a clinically significant abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product. Medical conditions present at baseline that worsened in severity or frequency after exposure to study drug were considered TEAEs. TEAEs were graded for severity (i.e., intensity) using Common Terminology Criteria for Adverse Events (CTCAE), version 5.0. Grade 1: mild; asymptomatic or mild symptoms; intervention not indicated. Grade 2: moderate; minimal, local or noninvasive intervention indicated. Grade 3: severe or medically significant, but not immediately life-threatening. Grade 4: life-threatening consequences; urgent intervention indicated. Grade 5: death related to TEAE.
Time Frame: up to 81 days
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | EP262 50 mg | EP262 150 mg
Number analyzed (Participants) | 38 | 37 | 38
Participants | 1 | 0 | 1

4. Secondary Outcome: Number of Participants With Any Clinically Meaningful Change From Baseline in Electrocardiogram Parameters
Description: Clinically meaningful changes were determined by the investigator.
Time Frame: up to 81 days
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | EP262 50 mg | EP262 150 mg
Number analyzed (Participants) | 38 | 37 | 38
Participants | 0 | 0 | 0

5. Secondary Outcome: Number of Participants With Any Clinically Meaningful Change From Baseline in Vital Sign Measurements
Description: Clinically meaningful changes were determined by the investigator.
Time Frame: up to 81 days
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | EP262 50 mg | EP262 150 mg
Number analyzed (Participants) | 38 | 37 | 38
Participants | 0 | 0 | 0

6. Secondary Outcome: Number of Participants With Any Clinically Meaningful Change From Baseline in Clinical Laboratory Test Results
Description: Clinically meaningful changes were determined by the investigator.
Time Frame: up to 81 days
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | EP262 50 mg | EP262 150 mg
Number analyzed (Participants) | 38 | 37 | 38
Participants | 4 | 4 | 5

7. Secondary Outcome: Change From Baseline to Visit 4 (Week 6) in the Itch Severity Score Over a 7-day Period (ISS7)
Description: The ISS is part of the UAS, a CSU-specific, 24-hour self-evaluation, patient-reported outcome measure based on the assessment of key CSU symptoms: intensity of itch (assessed as the ISS) and number of wheals (assessed as the HSS). The UAS scale for itch is recorded as a score from 0 to 3, with 0 representing no itch to 3 representing intense itch. ISS scores are summed over 7 consecutive days to create the ISS7 score, which ranges from 0 to 21. Higher scores indicate greater disease severity. The 7 daily ISS scores prior to or on the nominal Visit 4 (Week 6) date (including the nominal Week 6 visit date ISS score) were summed. Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline; Week 6
Population: Full Analysis Set. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo | EP262 50 mg | EP262 150 mg
Number analyzed (Participants) | 38 | 37 | 38
scores on a scale
  Baseline | 15.57 (3.918) | 13.55 (3.483) | 13.91 (4.016)
  Change from Baseline at Week 6: number analyzed (Participants) | 35 | 36 | 34
  Change from Baseline at Week 6 | -7.12 (6.058) | -4.89 (5.895) | -7.19 (5.631)

8. Secondary Outcome: Change From Baseline to Visit 4 (Week 6) in the Hive Severity Score Over a 7-day Period (HSS7)
Description: The HSS is part of the UAS, a CSU-specific, 24-hour self-evaluation, patient-reported outcome measure based on the assessment of key CSU symptoms: intensity of itch (assessed as the ISS) and number of wheals (assessed as the HSS). The UAS scale for wheal assessment is recorded as a score from 0 to 3, with 0 representing no hives to 3 representing intense hives. HSS scores are summed over 7 consecutive days to create the HSS7 score, which ranges from 0 to 21. Higher scores indicate greater disease severity. The 7 daily HSS scores prior to or on the nominal Visit 4 (Week 6) date (including the nominal Week 6 visit date HSS score) were summed. Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline; Week 6
Population: Full Analysis Set. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo | EP262 50 mg | EP262 150 mg
Number analyzed (Participants) | 38 | 37 | 38
scores on a scale
  Baseline | 13.95 (4.620) | 12.33 (4.331) | 12.04 (5.295)
  Change from Baseline at Week 6: number analyzed (Participants) | 35 | 36 | 34
  Change from Baseline at Week 6 | -5.71 (5.355) | -4.45 (5.584) | -5.66 (4.998)

ADVERSE EVENTS:
Time Frame: up to 81 days
Description: Adverse events have been reported for the Safety Analysis Set, comprised of all participants who were randomized and took at least 1 dose of randomized study drug.
Groups:
- EP262 Pooled: Participants received oral EP262 50 milligrams (mg) or 150 mg once daily for 6 weeks.
- EP262 50 mg: Participants received oral EP262 50 mg once daily for 6 weeks.
- Total: Total
Arm/Group | Placebo | EP262 Pooled | EP262 50 mg | EP262 150 mg | Total
All-Cause Mortality (participants affected / at risk) | 0/38 | 0/75 | 0/37 | 0/38 | 0/113
Serious Adverse Events (participants affected / at risk) | 0/38 | 0/75 | 0/37 | 0/38 | 0/113
Other Adverse Events (participants affected / at risk) | 6/38 | 14/75 | 6/37 | 8/38 | 20/113
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=38) | EP262 Pooled (N=75) | EP262 50 mg (N=37) | EP262 150 mg (N=38) | Total (N=113)
Blood creatine phosphokinase increased (Investigations) | 3 (3) | 2 (2) | 2 (2) | 0 (0) | 5 (5)
Bronchitis (Infections and infestations) | 0 (0) | 3 (3) | 1 (1) | 2 (2) | 3 (3)
Headache (Nervous system disorders) | 2 (3) | 3 (3) | 2 (2) | 1 (1) | 5 (6)
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 2 (2)
Nasopharyngitis (Infections and infestations) | 1 (1) | 3 (4) | 1 (2) | 2 (2) | 4 (5)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 2 (2)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 2 (2)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (3) | 0 (0) | 2 (3) | 2 (3)

LIMITATIONS AND CAVEATS:
The study was terminated following the completion of Part 1 due to business reasons; Part 2 was not enrolled.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 60 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.

DOCUMENTS (2):
  • Study Protocol (2024-07-26): https://cdn.clinicaltrials.gov/large-docs/73/NCT06077773/Prot_000.pdf
  • Statistical Analysis Plan (2025-01-31): https://cdn.clinicaltrials.gov/large-docs/73/NCT06077773/SAP_001.pdf